CLINICAL TRIAL: NCT02885948
Title: The NAPRESSIM Trial. The Use of Low Dose Prophylactic Naloxone Infusion to Prevent Respiratory Depression With Intrathecal Morphine.
Brief Title: The Use of Low Dose Prophylactic Naloxone Infusion to Prevent Respiratory Depression With Intrathecal Morphine.
Acronym: NAPRESSIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCDCRC/15/006
Record Dates: First submitted 2016-07-04; First posted 2016-09-01 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naloxone (Experimental): The naloxone arm of the study will receive naloxone at a rate of 5mcg/kg/hr which equates to 0.25ml/kg/hr. Each 1 ml ampoule of solution contains 400 micrograms (0.4mg) naloxone hydrochloride present as naloxone hydrochloride dihydrate.
  Excipients: each 1ml contains 3.55mg sodium. This will be diluted to a concentration of 20mcg/ml with 0.9% NaCl. Presented as solution for injection or infusion. Clear colourless sterile solution.
  Interventions: Drug: Naloxone
- Saline (Placebo Comparator): The placebo arm of the study will receive an infusion of normal saline at a rate of 0.25ml/kg/hr.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naloxone — used to block the effects of opioids, especially in overdose
  Arms: Naloxone
Drug: Placebo — Placebo, ineffective control arm
  Other Names: Placebo Saline
  Arms: Saline

SUMMARY:
This is an investigator led, randomised, double blind, placebo controlled, double arm comparator study.

DETAILED DESCRIPTION:
Delayed respiratory depression is a well-documented side effect associated with the use of intrathecal morphine. This respiratory depression has implications for patient safety and necessitates either the observation of the patient in a high dependency setting for at least 24 hours or the use of an alternative analgesic technique. Other associated side effects include pruritus, nausea and vomiting and sedation. Naloxone is the most effective treatment for these side effects. However, it is usually given as a reactive treatment when the side effect presents.

The hypothesis is that patients who are commenced on a naloxone infusion at low dose early after injection of intrathecal morphine will have a clinically significant reduction in incidence of these side effects. The primary endpoint is a reduction in respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be aged 18 years or above at baseline
* Diagnosed with any hepatobiliary condition requiring an elective major surgical resection under general anaesthetic.
* Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol

Exclusion Criteria:

* Allergy/sensitivity to naloxone
* Female subjects who are pregnant or breast-feeding.
* Subjects who have received any other investigational agent within 2 months
* Subjects taking anticonvulsant medications for epilepsy
* Subjects who have a cardiac arrhythmia with an uncontrolled rate
* Subjects who have a history of chronic opioid use / chronic pain
* Any contraindication to intrathecal injection eg coagulopathy
* Documented history of obstructive sleep apnoea
* Treating clinician feels not in the patients best interests to be randomised

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Respiratory depression | within 16 - 24 hours of participation

SECONDARY OUTCOMES:
Measure of occurrence of pain | within 16 - 24 hours of participation
Requirement for rescue analgesia | within 16 - 24 hours of participation
Nausea/Vomiting | within 16 - 24 hours of participation
Pruritus | within 16 - 24 hours of participation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Doran, PhD, Study Director — UCD
Locations (1):
- Prof. Alistair Nichol, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cosgrave D, Vencken S, Galligan M, McGuinness S, Soukhin E, McMullan V, Nair S, Puttappa A, Boylan J, Hussain R, Conlon N, Doran P, Nichol A. The effect of a low-dose naloxone infusion on the incidence of respiratory depression after intrathecal morphine administration for major open hepatobiliary surgery: a randomised controlled trial. Anaesthesia. 2020 Jun;75(6):747-755. doi: 10.1111/anae.14931. Epub 2019 Dec 2. PMID 31792949
- [Derived] Cosgrave D, Galligan M, Soukhin E, McMullan V, McGuinness S, Puttappa A, Conlon N, Boylan J, Hussain R, Doran P, Nichol A. The NAPRESSIM trial: the use of low-dose, prophylactic naloxone infusion to prevent respiratory depression with intrathecally administered morphine in elective hepatobiliary surgery: a study protocol and statistical analysis plan for a randomised controlled trial. Trials. 2017 Dec 29;18(1):633. doi: 10.1186/s13063-017-2370-0. PMID 29284510